CLINICAL TRIAL: NCT01844817
Title: A Randomized, Double-Blinded, Placebo-Controlled Phase II Trial Of Gemcitabine Plus Nab-Paclitaxel Combined With OGX-427 Or Placebo In Patients With Metastatic Pancreatic Cancer (The Rainier Trial)
Brief Title: Phase II Trial Of Gemcitabine Plus Nab-Paclitaxel +/- OGX-427 In Patients With Metastatic Pancreatic Cancer
Acronym: Rainier
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCRI GI 184
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: untreated; metastatic; OGX-427
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — apatorsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OGX-427 (Experimental): Three loading doses of OGX-427 at 600mg IV will be administered Days -9 to -1. Following the loading dose period, OGX-427 will be administered at 600mg IV weekly Days 1, 8, 15, and 22 of each 28 day cycle during the Treatment Phase.
  Interventions: Drug: OGX-427
- Placebo (Placebo Comparator): Three loading doses of placebo will be administered Days -9 to -1. Following the loading dose period, placebo will be administered weekly Days 1, 8, 15, and 22 of each 28 day cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OGX-427 — Three separate administrations of OGX-427 will be given during the 9-day Loading Dose Period. Following the Loading Dose Period, patients will receive 600mg OGX-427 prior to the administration of nab-paclitaxel (125mg/m2 IV)and gemcitabine (1000mg/m2 IV)administration on Day 1, 8, and 15 of each cycle. OGX-427 will also be administered on Day 22 during each cycle (i.e., weekly). Patients will continue 28 day treatment cycles until disease progression or until other reasons for discontinuation from treatment.
  Arms: OGX-427
Drug: Placebo — Three separate administrations of Placebo will be given during the 9-day Loading Dose Period. Following the Loading Dose Period, patients will receive placebo prior to the administration of nab-paclitaxel (125mg/m2 IV)and gemcitabine (1000mg/m2 IV)administration on Day 1, 8, and 15 of each cycle. Placebo will also be administered on Day 22 during each cycle (i.e., weekly). Patients will continue 28 day treatment cycles until disease progression or until other reasons for discontinuation from treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the overall survival in patients with previously untreated metastatic pancreatic cancer receiving gemcitabine/nab-paclitaxel plus OGX-427 or gemcitabine/nab-paclitaxel plus placebo.

DETAILED DESCRIPTION:
Patients with pancreatic cancer usually present with inoperable disease and systemic therapy becomes the primary form of treatment. The combination of gemcitabine plus nab-paclitaxel represents an appropriate front-line standard of care for patients with metastatic pancreatic cancer. However, poor outcomes with this disease warrant exploration of novel drugs with unique mechanisms of action. Preclinical evidence suggests that OGX-427 has shown promising activity in pancreatic cancer. In this trial, we will compare the overall survival of patients with previously untreated metastatic pancreatic cancer using OGX-427 with either gemcitabine/nab-paclitaxel or a placebo with gemcitabine/nab-paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically confirmed pancreatic adenocarcinoma
2. Stage IV disease (measurable disease NOT required)
3. Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
4. At least 18 years of age
5. Female patients who are not of child-bearing potential, and fertile female patients of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to start of randomization.
6. Fertile male patients willing to use adequate contraceptive measures.
7. Adequate bone marrow, renal, and hepatic function.
8. Ability to understand the nature of this study protocol, comply with study and/or follow-up procedures, and give written informed consent
9. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Any prior systemic or investigational therapy for metastatic pancreatic cancer. Systemic therapy administered alone or in combination with radiation in the adjuvant or neoadjuvant setting is permissible as long as it was completed > 6 months prior to the time of study randomization.
2. History of other diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
3. Presence of known central nervous system or brain metastases.
4. Known human immunodeficiency virus (HIV) infection.
5. Active second invasive malignancy (except non-melanomatous skin cancer), defined as any malignancy with current need for cancer therapy or high possibility (>30%) of recurrence during the study.
6. Patients receiving warfarin. However, therapeutic anticoagulation with Low Molecular Weight Heparin (LMWH) is allowed.
7. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease, and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months.
8. Current sensory neuropathy > Grade 1.
9. Major surgery within 4 weeks of the start of study treatment (defined as those surgeries that require general anesthesia. Insertion of a vascular access device is NOT considered major surgery.). Patients must have recovered from the side effects of any major surgery prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, M.D., Study Chair — SCRI
Locations (11):
- United States (11):
  - University of California-San Francisco, San Francisco, California
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Florida Hospital Cancer Insitute, Orlando, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Derived] Ko AH, Murphy PB, Peyton JD, Shipley DL, Al-Hazzouri A, Rodriguez FA, Womack MS 4th, Xiong HQ, Waterhouse DM, Tempero MA, Guo S, Lane CM, Earwood C, DeBusk LM, Bendell JC. A Randomized, Double-Blinded, Phase II Trial of Gemcitabine and Nab-Paclitaxel Plus Apatorsen or Placebo in Patients with Metastatic Pancreatic Cancer: The RAINIER Trial. Oncologist. 2017 Dec;22(12):1427-e129. doi: 10.1634/theoncologist.2017-0066. Epub 2017 Sep 21. PMID 28935773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2013 and December 2014, 132 subjhects with untreated metastatic pancreatic cancer were enrolled in the trial from 11 U.S. investigational sites.
Pre-assignment Details: Subjects were enrolled and randomized in a 1:1 ratio (66 per Arm) to receive a combination of gemcitabine and nab-paclitaxel plus either OGX-427 (apatorsen) or a placebo.
Groups:
- OGX-427: OGX-427: Three separate loading doses at 600mg IV over 1 week prior to Cycle 1 of chemotherapy, followed by 600mg IV once weekly on Days 1, 8, 15, and 22 of each 28 day cycle concurrent with chemotherapy.
  Chemotherapy: nab-paclitaxel (125mg/m^2 IV) and gemcitabine (1000mg/m^2 IV) on Days 1, 8, and 15 of each cycle. Patients continued 28 day treatment cycles until disease progression or until other reasons for discontinuation from treatment.
- Placebo: Placebo (dextrose 5% in water): Three separate loading doses administered over 1 week prior to Cycle 1 of chemotherapy, followed by weekly doses on Days 1, 8, 15, and 22 of each 28 day cycle concurrent with chemotherapy.
  Chemotherapy: nab-paclitaxel (125mg/m^2 IV) and gemcitabine (1000mg/m^2 IV) on Days 1, 8, and 15 of each cycle. Patients continued 28 day treatment cycles until disease progression or until other reasons for discontinuation from treatment.
Period: Enrolled and Randomized
Arm/Group | OGX-427 | Placebo
Started | 66 | 66
Completed (5 patients withdrew prior to treatment.) | 64 | 63
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Period: Treatment
Arm/Group | OGX-427 | Placebo
Started | 64 | 63
Completed | 0 | 0
Not Completed | 64 | 63
Not completed — Progressive Disease | 27 | 36
Not completed — Adverse Event | 17 | 9
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Death | 10 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population: All patients who met eligibility requirements and gave written informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | OGX-427 | Placebo | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Median (Full Range); unit: years] | 66.5 [39 to 82] | 65.5 [47 to 83] | 66 [39 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 37 | 38 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 56 | 61 | 117
  Black/African American | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival defined as the time, in months, from date of randomization until date of death or date last known alive whichever comes first, assessed up to 2 years.
Time Frame: Up to 2 years
Population: Includes Intent-to-Treat Population: all subjects enrolled and randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | OGX-427 | Placebo
Number analyzed (Participants) | 66 | 66
months | 5.3 [3.2 to 7.0] | 6.9 [5.8 to 9.3]

2. Secondary Outcome: Progression-Free Survival
Description: The time (in months) that patients are progression-free, assessed from date of randomization to date of first documented disease progression or date of death from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest (nadir) sum while on study (this includes the baseline sum if that is the smallest on study), or the appearance of one or more new lesions.
Time Frame: Every 8 weeks up to 2 years
Population: Intent-to-Treat Population: all subjects enrolled and randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | OGX-427 | Placebo
Number analyzed (Participants) | 66 | 66
months | 2.7 [2.2 to 3.7] | 3.8 [2.3 to 4.7]

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate defined as the percent of patients having a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR=complete disappearance of all target lesions. PR=decrease in baseline of 30% or more of the diameter(s) of all target lesions.
Time Frame: Every 8 weeks for up to 2 years
Population: Includes Intent-to-Treat Population: all subjects enrolled and randomized
Measure: Number; unit: percentage of participants
Arm/Group | OGX-427 | Placebo
Number analyzed (Participants) | 66 | 66
percentage of participants
  PR | 18 | 18
  CR | 0 | 0

ADVERSE EVENTS:
Time Frame: weekly for approximately 24 months
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from day of first dose to 30 days after last dose of study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | OGX-427 | Placebo
Serious Adverse Events (participants affected / at risk) | 64/64 | 63/63
Other Adverse Events (participants affected / at risk) | 62/64 | 62/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-427 (N=64) | Placebo (N=63)
Dehydration (Metabolism and nutrition disorders) | 18 | 12
Sepsis (Infections and infestations) | 18 | 9
Abdominal Pain (Gastrointestinal disorders) | 12 | 9
Pneumonia (Infections and infestations) | 12 | 6
Acute Kidney Injury (Renal and urinary disorders) | 12 | 3
Anaemia (Blood and lymphatic system disorders) | 9 | 6
Atrial Fibrillation (Cardiac disorders) | 9 | 6
Bile Duct Obstruction (Hepatobiliary disorders) | 9 | 3
Deep Vein Thrombosis (Vascular disorders) | 3 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 9 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pyrexia (General disorders) | 12 | 0
Cellulitis (Infections and infestations) | 3 | 6
Obstruction Gastric (Gastrointestinal disorders) | 0 | 9
Vomiting (Gastrointestinal disorders) | 3 | 6
Acute Myocardial Infarction (Cardiac disorders) | 3 | 3
Cardiac Failure Congestive (Cardiac disorders) | 0 | 6
Cerebrovascular Accident (Vascular disorders) | 6 | 0
Device Occlusion (General disorders) | 0 | 6
Fatigue (General disorders) | 6 | 0
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 3
Renal Failure (Renal and urinary disorders) | 3 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Small Intestine Obstruction (Hepatobiliary disorders) | 3 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0
Anaphylactic Reaction (Immune system disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 0 | 3
Asthenia (General disorders) | 0 | 3
Bacteraemia (Skin and subcutaneous tissue disorders) | 0 | 3
Biliary Tract Infection (Hepatobiliary disorders) | 0 | 3
Bursitis Infective Staphylococcal (Infections and infestations) | 0 | 3
Cardiac Arrest (Cardiac disorders) | 0 | 3
Chest Pain (General disorders) | 3 | 0
Cholangitis Infective (Infections and infestations) | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3
Device Related Infection (General disorders) | 0 | 3
Duodenal Obstruction (Gastrointestinal disorders) | 3 | 0
Duodenal Stenosis (Gastrointestinal disorders) | 3 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 3
Failure to Thrive (Investigations) | 0 | 3
Febrile Neutropeniua (Blood and lymphatic system disorders) | 0 | 3
Gastric Varices Haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastritis (Gastrointestinal disorders) | 3 | 0
Gastritis Erosive (Gastrointestinal disorders) | 3 | 0
Haematochezia (Hepatobiliary disorders) | 0 | 3
Haemorrhagic Ascites (Gastrointestinal disorders) | 0 | 3
Hypotension (Blood and lymphatic system disorders) | 0 | 3
Ileus Spastic (Gastrointestinal disorders) | 0 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 3
Ischaemic Stroke (Vascular disorders) | 3 | 0
Klebsiella Infection (Infections and infestations) | 3 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 3 | 0
Lethargy (General disorders) | 3 | 0
Mucosal Inflammation (General disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Oedema Peripheral (Nervous system disorders) | 3 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 3
Peptic Ulcer (Gastrointestinal disorders) | 3 | 0
Systemic Inflammatory Response (Nervous system disorders) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3
Urosepsis (Renal and urinary disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-427 (N=64) | Placebo (N=63)
Anaemia (Blood and lymphatic system disorders) | 36 | 40
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 21
Neutropenia (Blood and lymphatic system disorders) | 18 | 21
Leukopenia (Blood and lymphatic system disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 34 | 40
Abdominal Pain (Gastrointestinal disorders) | 26 | 21
Diarrhoea (Gastrointestinal disorders) | 28 | 18
Vomiting (Gastrointestinal disorders) | 26 | 20
Constipation (Gastrointestinal disorders) | 20 | 22
Dyspepsia (Gastrointestinal disorders) | 7 | 5
Ascites (Gastrointestinal disorders) | 5 | 5
Flatulence (Gastrointestinal disorders) | 4 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 2
Stomatitis (Gastrointestinal disorders) | 6 | 3
Gastroesophageal Reflux (Gastrointestinal disorders) | 4 | 4
Abdominal Distention (Gastrointestinal disorders) | 3 | 4
Fatigure (General disorders) | 41 | 44
Oedema Peripheral (General disorders) | 26 | 16
Pyrexia (General disorders) | 21 | 17
Asthenia (General disorders) | 9 | 11
Chills (General disorders) | 4 | 9
Pain (General disorders) | 5 | 4
Peripheral Swelling (General disorders) | 2 | 7
Mucosal Inflammation (General disorders) | 4 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 23 | 22
Dehydration (Metabolism and nutrition disorders) | 16 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5
Hyperalbuminaemia (Metabolism and nutrition disorders) | 4 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 3
Alanine Aminotransferase Increased (Investigations) | 16 | 16
Aspartate Aminotransferase Increased (Investigations) | 16 | 13
Platelet Count Decreased (Investigations) | 16 | 11
Blood Alkaline Phosphatase Increased (Investigations) | 11 | 13
Weight Decreased (Investigations) | 12 | 12
Neutrophil Count Decreased (Investigations) | 6 | 9
Blood Bilirubin Increased (Investigations) | 7 | 7
Blood Creatinine Increased (Investigations) | 8 | 4
Urinary Tract Infections (Infections and infestations) | 9 | 4
Pneumonia (Infections and infestations) | 6 | 3
Sepsis (Infections and infestations) | 5 | 4
Upper Respiratory Track Infection (Infections and infestations) | 6 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 15
Rash (Skin and subcutaneous tissue disorders) | 9 | 16
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 10 | 15
Anxiety (Psychiatric disorders) | 7 | 8
Depression (Psychiatric disorders) | 8 | 2
Hypotension (Vascular disorders) | 8 | 10
Deep Vein Thrombosis (Vascular disorders) | 4 | 8
Hypertension (Vascular disorders) | 4 | 7
Flushing (Vascular disorders) | 4 | 5
Acute Kidney Injury (Renal and urinary disorders) | 6 | 3
Tachycardia (Cardiac disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.